CLINICAL TRIAL: NCT02576405
Title: Characterization of Preoperative Psychiatric Disorder in Relation to Postoperative Morbidity in Elective Fast-Track Total Hip and Knee Arthroplasty
Brief Title: Psychiatric Disorder and Postoperative Morbidity in Hip and Knee Artroplasty
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Silas Hinsch Gylvin, Medical Doctor, Rigshospitalet, Denmark
Other Study IDs: SG
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-09

CONDITIONS: Focus is on Preoperative Psychiatric Charactarization of Elective Fast-track Hip and Knee Arthroplasty Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
It has been established that patients with psychiatric disorders tend to do worse in a surgical setting. Some types of surgery with greater impact than others, including orthopedic surgery. In our research group the investigators have shown this to be the case for hip and knee replacements within the mentioned patient category. However, the role of psychiatric disorder and use of different psychopharmacological drugs in relation to perioperative morbidity and mortality have not been thoroughly examined. The objective of this study is to shed light on the issue.

Recent studies have shown that different types of psychiatric disorder influence surgical outcome differently. This emphasizes the need for specific knowledge regarding psychiatric diagnoses preoperatively. In this study around 2000 patients with or without psychiatric disorder of any kind will be studied preoperatively, which according to our previous study will include more than 200 patients receiving psychopharmacological treatment. The specifics that characterize every patient's psychiatric trades will be included in a validated questionnaire constructed for that purpose. The questionnaire is called SCL-92 and has been chosen in collaboration with Professor in Psychiatry, Rigshospitalet Anders Fink-Jensen. Preoperative information regarding their mental condition and medicine will be linked to surgical outcome in order to identify potential hazards in the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* All patients planned for elective unilateral fast-track hip or knee arthroplasty.
* Age > 18.
* Can understand and read danish.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Danish population sample (N=2000) of hip and knee arthroplasty patients in an elective fast-track setting.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Psychological characterization of hip and knee arthroplasty patients using the validated SCL-92 questionnaire | 90 days postoperatively

SECONDARY OUTCOMES:
Length of stay | 90 days postoperatively
Readmissions | 30 and 90 days postoperatively